CLINICAL TRIAL: NCT03589339
Title: A Phase I Dose Escalation / Dose Expansion Study of NBTXR3 Activated by Radiotherapy for Patients With Advanced Cancers Treated With An Anti-PD-1 Therapy
Brief Title: NBTXR3 Activated by Radiotherapy for Patients With Advanced Cancers Treated With An Anti-PD-1 Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanobiotix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1100
Record Dates: First submitted 2018-04-10; First posted 2018-07-17 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Radiotherapy; Immunotherapy; Microsatellite Instability-High Solid Malignant Tumour; Metastasis From Malignant Tumor of Liver; Squamous Cell Carcinoma of Head and Neck; Metastasis From Malignant Tumor of Cervix; Metastatic Renal Cell Carcinoma; Metastasis From Malignant Melanoma of Skin (Disorder); Metastatic Triple-Negative Breast Carcinoma; Metastatic NSCLC; Metastasis From Malignant Tumor of Bladder (Disorder)
Keywords: Oral Cavity Cancer; Oropharynx Cancer; Lung Metastasis; Liver Metastasis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Mouth Neoplasms; Oropharyngeal Neoplasms | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBTXR3 activated by SABR followed by anti-PD-1 monotherapy (Experimental): Intratumoral injection of NBTXR3 followed by SABR followed by monotherapy with nivolumab or pembrolizumab
  Interventions: Drug: NBTXR3; Radiation: SABR; Drug: Nivolumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: NBTXR3 — Single intra Tumoral injection
Radiation: SABR — Radiotherapy given as a definite number of fractions at the dose defined for each radiation field
  Other Names: Stereotaxic Ablative Radiotherapy; Stereotaxic Body Radiation Therapy
Drug: Nivolumab — Anti-PD-1 monotherapy
  Other Names: Opdivo
Drug: Pembrolizumab — Anti-PD-1 monotherapy
  Other Names: Keytruda

SUMMARY:
The 1100 study is an open-label, Phase I, dose escalation and expansion prospective clinical study to assess the safety of intratumoral injection of NBTXR3 activated by radiotherapy in combination with anti-PD-1 therapy.

DETAILED DESCRIPTION:
The 1100 study aims to evaluate the safety, efficacy, and tolerability of NBTXR3 activated by radiotherapy in combination with an anti-PD-1 therapy in three cohorts of patients in dose escalation and expansion parts. The Escalation Cohort 1 includes patients with LRR or R/M HNSCC with the injectable lesion in a previously irradiated field. In Escalation Cohorts 2 and 3, patients present with lung or liver metastases from any primary cancer eligible for anti-PD-1 therapy.

The Expansion cohort 1 includes patients with LRR or R/M HNSCC with the injectable lesion located either in head and neck area or in lung or liver, who are resistant to anti-PD-1 therapy. The Expansion cohort 2 includes patients with LRR or R/M HNSCC with the injectable lesion located either in head and neck area or in lung or liver, who are naive to anti-PD-1 therapy.

The Expansion Cohort 3 includes patients with inoperable NSCLC, malignant melanoma, HCC, RCC, urothelial cancer, cervical cancer or TNBC with metastases to lungs, liver or soft tissue and who are resistant to anti-PD-1 therapy.

These patients have a high unmet need and the Sponsor hypothesizes that NBTXR3 activated by radiotherapy will act synergistically with anti-PD-1 to enhance the therapeutic index of radiotherapy maximizing local effect, to overcome radio-resistance, to increase the local efficacy of immunotherapy, and to improve distant tumor control via an abscopal effect. Eligible patients will receive a single intratumoral injection of NBTXR3 subsequently activated by radiotherapy and then an approved anti-PD-1. The end of treatment visit will take place 4 weeks after the last radiotherapy fraction. Patients will be followed for long-term safety and efficacy for 2 years after the EOT visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Biopsy-confirmed cancer diagnosis indicated to receive anti-PD-1 therapy:

Dose Escalation:

1. Escalation Cohort 1: Is inoperable LRR with tumor in previously irradiated HN field that is amenable to re-irradiation or R/M HNSCC with tumor in previously irradiated HN field that is amenable to re-irradiation, or
2. Escalation Cohort 2: Has metastasized to the lung (including involved lymph nodes) with tumor in a previously non-irradiated lung field, or
3. Escalation Cohort 3: Has metastasized to the liver with tumor in a previously non-irradiated liver field

Expansion:

1. Expansion Cohorts 1 and 2: Is inoperable LRR or R/M HNSCC with at least one lesion that is amenable to irradiation within head and neck region, lung or liver
2. Expansion Cohort 3: Is inoperable NSCLC, malignant melanoma, HCC, RCC, urothelial cancer, cervical cancer, TNBC that has metastasized to soft tissues, lung (including mediastinal lymph nodes) or liver with at least one lesion that is amenable to irradiation

   * Prior anti-PD-1 exposure as follows:

Dose Escalation (all cohorts):

1. Has not received prior anti-PD-1 therapy (i.e., anti-PD-1 naïve), or
2. Has received prior anti-PD-1 therapy and meets criteria consistent with anti-PD-1 primary resistance (i.e., primary anti-PD-1 non-responder), or
3. Has received prior anti-PD-1 therapy and meets criteria consistent with anti-PD-1 secondary resistance (i.e., secondary anti-PD-1 non-responder)

Expansion:

1. Expansion Cohorts 1 and 3: Has received prior anti-PD-1 therapy and meets criteria consistent with anti-PD-1 primary or secondary resistance as described above
2. Expansion Cohort 2: Has not received prior anti-PD-1 therapy (i.e., anti-PD-1 naïve)

   * Has at least one tumor lesion that can be accurately measured according to RECIST 1.1. and is amenable for intratumoral injection
   * ECOG performance status 0-2
   * Life expectancy >12 weeks
   * Adequate organ and bone marrow function
   * Negative pregnancy test ≤ 7 days prior to NBTXR3 injection in all female participants of child-bearing potential

Exclusion Criteria:

* History of immune-related adverse events related to administration of anti-PD-1/L1 that led to the termination of the previous anti-PD-1 therapy due to intolerance or toxicity and precludes further PD-1 exposure
* Symptomatic central nervous system metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 1 year
* Known HIV or active hepatitis B/C infection
* Active infection requiring intravenous treatment with antibiotics
* Received a live virus vaccine within 30 days prior to study treatment
* History of pneumonitis that required steroids or with current pneumonitis
* Extensive metastatic disease burden defined as more than 5 lesions overall including the primary tumor
* Locoregional recurrent HNSCC with ulceration
* Has received prior therapy with a checkpoint inhibitor, within 2 weeks prior to NBTXR3 injection
* Has received prior systemic anti-neoplastic therapy, including investigational agents, within 4 weeks prior to NBTXR3 injection
* Has not recovered from AEs due to previous anti-neoplastic therapies and/or interventions (including radiation) to ≤ Grade 1 or baseline at screening
* Clinically significant cardiac arrhythmias
* Class III or IV Congestive Heart Failure as defined by the New York Heart Association functional classification system < 6 months prior to screening
* A pregnant or nursing female, or women of child-bearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Any condition for which participation would not be in the best interest of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
[Dose Escalation Part]: Determination of the Recommended Dose | 24 Months
  Determination of DLTs, the MTD (if possible), and RP2Ds for each cohort
[Dose Expansion Part]: Safety Evaluation at RP2D | 24 Months
  Incidence of Grade 3 and higher treatment-related AEs

SECONDARY OUTCOMES:
Evaluation of the anti-tumor response of R3/RT/PD-1 | 24 months
  Evaluation of the Objective Response Rate: complete or partial response, as defined by RECIST 1.1 and iRECIST
Assessment of the safety and feasibility of R3/RT/PD-1 | 24 months
  Assessment of the number of participants with related late onset toxicities defined as any Grade ≥3 AE occurring after the EOT visit and determination of the number of participants with feasible NBTXR3 intratumoral injection
Evaluation of the body kinetic profile of intratumorally injected NBTXR3 | 24 months
  Evaluation of the time-course dependent accumulation of hafnium in blood and urine following NBTXR3 intratumoral injection

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Tyan, MD, Study Director — Nanobiotix
Locations (13):
- United States (13):
  - University of California San Francisco, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Christus St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Northwell Health, Manhasset, New York
  - University of North Carolina, School of Medicine, Chapel Hill, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - St Luke's University Health Network, Bethlehem, Pennsylvania
  - Sanford Cancer Center, Sioux Falls, South Dakota

REFERENCES:
- [Background] Shen C, Frakes J, Niu J, et al 684 NBTXR3 activated by radiotherapy in combination with nivolumab or pembrolizumab in patients with advanced cancers: results from an ongoing dose escalation phase I trial (Study 1100). Journal for ImmunoTherapy of Cancer 2022;10:doi: 10.1136/jitc-2022-SITC2022.0684